CLINICAL TRIAL: NCT02221726
Title: Evaluation of Scoring Methods to Assess Adhesion Quality and Wear of the Placebo JNJ-35685-AAA-G-023 5.5 cm^2 and 44 cm^2 Transdermal Systems
Brief Title: Study to Assess Adhesion Quality and Wear of Placebo JNJ-35685-AAA-G-023 Transdermal System in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105188; FENPAI1024 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy; JNJ-35685-AAA-G-023; Placebo; Transdermal delivery device system

ARMS (2):
- JNJ-35684-AAA-023: 5.5 cm^2 Patch (Experimental)
  Interventions: Drug: JNJ-35684-AAA-023: Size 1; small patch
- JNJ-35684-AAA-023: 44 cm^2 Patch (Experimental)
  Interventions: Drug: JNJ-35684-AAA-023: Size 2; large patch

INTERVENTIONS:
Drug: JNJ-35684-AAA-023: Size 1; small patch — Placebo (matched to Fentanyl transdermal delivery device system [TDDS]) JNJ-35685-AAA-G-023 TDDS, 5.5 centimeter square (cm^2) will be applied vertically to 1 side of the paraspinal region, replicated 3 times, and worn for 72 hours.
  Arms: JNJ-35684-AAA-023: 5.5 cm^2 Patch
Drug: JNJ-35684-AAA-023: Size 2; large patch — Placebo (matched to Fentanyl transdermal delivery device system [TDDS]) JNJ-35685-AAA-G-023 TDDS, 44 cm^2 (Size 1; small patch) will be applied vertically to other side of the paraspinal region, replicated 3 times, and worn for 72 hours.
  Arms: JNJ-35684-AAA-023: 44 cm^2 Patch

SUMMARY:
The purpose of this study is to assess 3 different scoring systems to evaluate the adhesive quality of placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial]) JNJ-35685-AAA-G-023-G transdermal (through the skin) systems during a single system 72-hour application, replicated 3 times, of 2 patch sizes (5.5 centimeter^2 [cm^2] and 44 cm^2).

DETAILED DESCRIPTION:
This study will assess 3 different scoring systems to evaluate the adhesive quality of "placebo" patch (an inactive patch that contains no active drug), JNJ-35685-AAA-G-023-G transdermal (through the skin) system. In this study, this patch is NOT being compared to a patch with a drug, and is NOT being used to test if the patch with the drug has a real effect in a clinical trial. The study consists 3 parts: Screening (21 days before study commences on Day 1), an adhesion assessment period (4 days), and an end of Study (EOS) assessment (recorded at 24 hours +/- 4 hours following patch removal). Total study duration per participant will be 26 days (including Screening). JNJ-35685-AAA-G-023 small (5.5 cm^2) and large (44 cm^2) patches will be applied on to left or right side of the paraspinal region based on randomization schedule. Adhesion assessments will be performed at patch application (hour 0, Baseline), and during the time interval of 8 to 10 hours, 24, 48, and 72 hours following patch application. Adhesion quality will be assessed by visual grading, United States Food and Drug Administration (FDA) scale, digital image analysis and visual grading grid system. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI: weight in kilogram [kg]/height^2 [meter (m^2)]) between 18 and 35 kg/m^2 (inclusive), and body weight not less than 50 kg
* Blood pressure (can be taken in supine or sitting position) between 90 and 140 milimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker (for at least 6 months prior to screening) and willing to abstain from smoking during the study confinement period
* Good general health as determined by medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests
* Willing to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* History of or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); lipid abnormalities; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal insufficiency (creatinine clearance below 60 milliliter per minute [mL/min]); thyroid disease; neurologic or psychiatric disease; infection; or any other illness that the Investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the Investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening as deemed appropriate by the Investigator
* Use of medications or treatments that would significantly influence or exaggerate patch adhesion or that would alter inflammatory or immune response to the study product (example, antihistamines, systemic or topical corticosteroids, cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin (BCG), monoclonal antibodies, radiation therapy)
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Visual Grading United States Food and Drug Administration (FDA) Scale Score | Baseline up to 72 hours following patch application
  Visual grading US FDA scale will be used to evaluate adhesion performance of the transdermal system. The score ranges from 0-4: 0 = greater than or equal to (>=) 90 percent (%) adhered (essentially no lift off the skin); 1 = greater than or equal to 75% to less than (<) 90% adhered (some edges only lifting off the skin); 2 = greater than or equal to 50% to <75% adhered (less than half of the patch lifting off the skin); 3 = greater than (>) 0% to <50% adhered but not detached (more than half of the patch lifting off the skin without falling off); and 4 = 0% adhered - patch detached (patch completely off the skin).
Adhesion Area Calculated by Digital Image Analysis | Baseline up to 72 hours following patch application
  Digital image will be captured with high resolution for each transdermal patch site and adhesion area will be calculated.
Total Adhesion Score Calculated by Visual Grading Grid System | Baseline up to 72 hours following patch application
  Total adhesion score will be calculated by visual grading grid system (a grid system based on 20 four-sided divisions that are approximately 5% of the total patch area; 44 cm^2 patch will be evaluated by square and rectangular grid elements while 5.5 cm^2 patch will be evaluated by square grid element only) which also contains a scale to allow for proper determination of actual area of the patch not adhering to the skin. Total area of the patch which does not adhere will be calculated. Any area of the patch that does not entirely adhere onto the skin will be scored as 0% adhesion for that area. Subsequently, a total adhesion score for that system will be calculated.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs | Baseline up to 72 hours following patch application

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States